CLINICAL TRIAL: NCT05549791
Title: A Domestic, Prospective, Non-interventional Study of Remimazolam Tosilate for Injection in the Real-world for General Anesthesia and Fiberoptic Bronchoscopy Sedation
Brief Title: A Non-intervention Fiberoptic Bronchoscopy Study of Remazolam Toluene Sulfonate for Injection Under General Anesthesia and Fiberoptic Bronchoscopy
Status: Completed | Type: Observational
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: ARMS-
Record Dates: First submitted 2022-08-24; First posted 2022-09-22 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: General Anesthesia and Bronchoscopy Sedation
MeSH Terms: interventions — Injections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General anesthesia cohort
  Interventions: Drug: Remimazolam Tosilate for Injection
- Bronchoscopy sedation cohort
  Interventions: Drug: Remimazolam Tosilate for Injection

INTERVENTIONS:
Drug: Remimazolam Tosilate for Injection — Remimazolam Tosilate for Injection

SUMMARY:
This is a non-interventional study of remazolam toluenesulfonate (rebenin ®) for injection in Chinese patients. A total of 1000 patients were enrolled in this study based on the preliminary safety assessment of rebenin ®, and all safety information was obtained

ELIGIBILITY:
Inclusion Criteria:

1. Patients using rebinim ® during general anesthesia and fiberoptic sedation
2. Patients need to sign informed consent

Exclusion Criteria:

1. Patients who are participating in or planning to participate in any interventional clinical trial
2. The investigator considers that there are any other reasons for the patient's ineligibility for the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients receiving remazolam toluenesulfonate for general anesthesia or bronchoscopy sedation
Sampling Method: Non-Probability Sample
Enrollment: 1285 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-21 (Actual)

PRIMARY OUTCOMES:
Adverse events | Within 3 days of receiving General anesthesia and bronchoscopy sedation
  Use adverse event record form,Refer to version 5.0 of the NCI-CTCAE

SECONDARY OUTCOMES:
Serious adverse events | Within 3 days of receiving General anesthesia and bronchoscopy sedation
  Refer to SAE definition standards
Adverse drug reactions | Within 3 days of receiving General anesthesia and bronchoscopy sedation
  By evaluating the association of adverse events with drugs
Injection pain | Within 3 days of receiving General anesthesia and bronchoscopy sedation
  Refer to the NCI-CTCAE <5.0> grading criteria for drug injection site reactions

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided